CLINICAL TRIAL: NCT01770886
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral UE2343 in Healthy Subjects
Brief Title: A Phase I Study of Oral UE2343 in Healthy Subjects
Acronym: UE2343
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Wellcome Trust (Other); Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UE2343
Record Dates: First submitted 2013-01-10; First posted 2013-01-18 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Drug Safety
MeSH Terms: interventions — UE2343

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UE2343 (Active Comparator): Oral capsule
  Interventions: Drug: UE2343
- Placebo (Placebo Comparator): Oral capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UE2343 — Oral capsule
  Arms: UE2343
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
A randomised, double-blind, placebo-controlled, phase I study in healthy subjects. Safety, pharmacokinetic and pharmacodynamic data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 and 65 years of age (inclusive).
* Female subject is postmenopausal or surgically sterilized or had a hysterectomy.
* Female subject with negative pregnancy test.
* Male subjects willing to use an effective method of contraception, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from Day 1 until 3 months afterwards.
* Subject with a Body Mass Index (BMI) of 18-30 kg/m2. Body Mass Index = Body weight (kg) / [Height (m)]2.
* Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values or results suggesting an infectious or other systemic disorder. The parameters to be measured will include those shown in Appendix 2. The Simbec normal ranges are shown in Appendix 3.
* Subject with a negative urinary drugs of abuse screen (Appendix 2) (N.B. a positive alcohol result may be repeated at the discretion of the Investigator).
* Subject with negative HIV and Hepatitis B and C results.
* Subject with no clinically significant abnormalities in 12-lead electrocardiogram (ECG).
* no clinically significant abnormalities in vital signs.
* willing and able to comply with the requirements of the protocol.
* satisfy a medical examiner about fitness to participate in the study.
* provide written informed consent to participate in the study.
* Smokers are eligible to participate in the study.

Exclusion Criteria:

* Relevant abnormality in medical history or on examination, including history of dementia, or other psychiatric, neurological, immunological, respiratory or cardiovascular disorder. Particularly exclude subjects with signs of peripheral neuropathy. Abnormal laboratory findings suggesting the presence of a systematic disorder.
* Participation in a clinical study of an unlicensed drug in the previous 4 months, or a marketed drug study within the previous 3 months. (N.B. washout period between trials defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
* Known allergies, including allergy to chemicals like and excipients associated with UE2343.
* Recent or clinically significant history of drug or alcohol abuse.
* Blood donation greater than 500 ml in the previous 3 months.
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Receipt of regular prescribed medication within 7 days of the first study day and / or receipt of vitamins, minerals, herbal remedies and nutritional supplements within 7 days of the first study day. Subjects taking long lasting drugs more than 7 days before the study may be excluded at the physician's discretion. Inclusion of subjects who have taken over the counter drugs during this period will be reviewed on a case-by-case basis in relation to the safety aspects and objectives of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of UE2343 in healthy male/female subjects | At each dose
  Days 1-2 at each dose:
  * 12 lead ECG
  * Vital signs
  * Symptom led clinical assessment (day 1 only)
  * Routine laboratory assessments
  Days 3-6 at each dose:
  * 12 lead ECG
  * Vital signs
  * Routine laboratory assessments
  Day 10 at each dose:
  * 12 lead ECG
  * Vital signs
  * Routine laboratory assessments
  * Physical examination
  * Pregnancy test

SECONDARY OUTCOMES:
Pharmacokinetic parameters of UE2343 and pharmacodynamic exposure | At each dose
  Days 1-2 at each dose:
  * Blood and urine samples for measurement of UE2343
  * Blood samples for adrenal androgens
  * Blood samples for ACTH and cortisol
  * Urine samples for urinary free steroids
  Days 3-6 at each dose:
  * Blood and urine samples for measurement of UE2343
  * Blood samples for adrenal androgens
  * Blood samples for ACTH and cortisol
  * Urine samples for urinary free steroids

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Walker, BSc MBChB MD, Principal Investigator — University of Edinburgh
Locations (1):
- Simbec Research, Merthyr Tydfil, United Kingdom